CLINICAL TRIAL: NCT05782478
Title: Added Diagnostic Value of Point of Care Ultrasound in Acute Dyspnea: a Prospective Observational Study
Brief Title: Added Diagnostic Value of Point of Care Ultrasound in Acute Dyspnea
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02789-01
Record Dates: First submitted 2023-03-08; First posted 2023-03-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Dyspnea; Hypoxia
Keywords: Ultrasound; Point of care ultrasound
MeSH Terms: conditions — Dyspnea; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Point of care Ultrasound according to study protocol — An emergency medicine specialist or resident will according to a structured protocol perform a structured ultrasound examination of the heart, the inferior vena cava and the lungs.

SUMMARY:
Dyspnea is a common diagnostic challenge in the Emergency Department (ED). Delay in diagnosis will increase time to correct treatment and could impact outcome. Previous studies have shown excellent diagnostic performance of point of care ultrasound (POCUS) to detect and differentiate between several important diagnosis (e.g heart failure and pneumonia) in patients with dyspnea. However, in most studies POCUS is performed by physicians highly experienced in ultrasound and often studies have focused only on one or few diagnoses. The aim of this study is to compare the diagnostic accuracy of different diagnosis in dyspnoeic patients before and after a ED physician with limited training applies POCUS.

DETAILED DESCRIPTION:
Dyspnoea is a common presenting complaint in the Emergency Department (ED). Dyspnoea requires timely evaluation and treatment as several conditions causing dyspnea are time critical.

Previous studies have suggested that point-of-care ultrasound (POCUS) increase diagnostic accuracy in the initial assessment of patients with dyspnoea. However, in most studies POCUS was done by highly experienced physicians which could limit the generalisability of POCUS in the hands of all emergency specialist and residents.

Aim To evaluate whether POCUS performed by a variety of emergency medicine physicians (specialists and residents) increase diagnostic accuracy in patients with dyspnea compared to routine assessment.

Method:

Specialist and residents in Emergency Medicine at the ED in Lund and Helsingborg (Sweden) will have a short training and certification in a structured dyspnea POCUS protocol. The protocol includes focused lung (8 or 14 zones), heart (subcostal, parasternal and apical four chamber views) and inferior vena cava ultrasound.

Study design Prospective observational study

Study population

Inclusion criteria

Adult patients presenting to the Emergency Department within the highest or second highest triage category (Rapid Emergency Triage and Treatment System) and any of the following:

* Presenting with shortness of breath
* Oxygen saturation less than 90 % on room air
* Respiratory rate more than 25 breaths per minute and oxygen saturation less than 95 % on room air

Exclusion criteria

* Inclusion in the study will delay urgent interventions
* Patient is discharge from the ED (without hospital admission)

Patients will be included when a physician certified in the dyspnea POUCUS protocol is present in the ED (convenience sample) Firstly, an ED physician will assess the patient using available routine diagnostic procedures. After consent to the study, the physician will document the estimated likelihood (not likely, unlikely, likely, very likely) of the following diagnosis: heart failure, pulmonary embolism, pneumonia, exacerbation of chronic obstructive pulmonary disease (COPD), exacerbation of asthma, pleural or pericardial fluid. Clinical bedside tests will be available as in routine practice in the ED (e.g., ecg, blood gas results). A physician certified in the dyspnea protocol will then perform POCUS and deliver the findings to the initial physician assessing the patients. Hereafter, the initial physician documents the estimated likelihood of the above diagnosis being provided the ultrasound findings.

The estimated likelihoods (before and after POCUS) will be dichotomised and compared to the discharge diagnosis. Sensitivity, specificity, negative and positive predictive values of the diagnostic accuracy before and after adding POCUS will be calculated.

In addition to routine bed-side tests alle included patients will have the following ordered: chest imaging (x-ray or CT according to ED physicians' choice), N-terminal pro-B-type natriuretic peptide (pro-BNP), C-reactive protein and white blood count.

ELIGIBILITY:
Inclusion Criteria:

Adult patients presenting to the Emergency Department within the highest or second highest triage category and any of the following

* Presenting with shortness of breath
* Oxygen saturation less than 90 % on room air
* Respiratory rate more than 25 breaths per minute and oxygen saturation less than 95 % on room air

Exclusion Criteria:

* Inclusion in the study will delay urgent interventions
* Patient is discharge from the Emergency Department (without hospital admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Department at Skåne University Hospital in Lund or Helsingborg Hospital, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Discharge diagnosis | Final diagnosis at index visit discharge
  Any of the following diagnosis: Decompensated heart failure, pulmonary embolism, COPD exacerbation, asthma exacerbation, bacterial pneumonia, viral pneumonia, pleural fluid, pericardial fluid

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lundager Forberg, PhD,MD, Principal Investigator — Region Skåne Sweden
Locations (2):
- Sweden (2):
  - Department of Emergency Medicine, Helsingborg Hospital, Helsingborg, Skåne County
  - Department of Emergency Medicine, Skåne University Hospital, Lund, Skåne County